CLINICAL TRIAL: NCT02781480
Title: An Open-label, Multi-centre, Phase I/II Dose Escalation Trial of an Adeno Associated Virus Vector for Gene Therapy of Adults And Children With Retinal Dystrophy Associated With Defects in RPE65 (LCA)
Brief Title: Clinical Trial of Gene Therapy for the Treatment of Leber Congenital Amaurosis (LCA)
Acronym: OPTIRPE65
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MeiraGTx UK II Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MGT003
Record Dates: First submitted 2016-04-28; First posted 2016-05-24 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Leber Congenital Amaurosis
MeSH Terms: conditions — Leber Congenital Amaurosis

STUDY DESIGN:
Intervention Model Description: AAV2/5-OPTIRPE65
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose AAV-RPE65 (Experimental): Subretinal administration of a single low dose of range AAV-RPE65
  Interventions: Biological: AAV RPE65
- Intermediate dose AAV-RPE65 (Experimental): Subretinal administration of a single intermediate dose of range AAV-RPE65
  Interventions: Biological: AAV RPE65
- High dose AAV-RPE65 (Experimental): Subretinal administration of a single high dose of range AAV-RPE65
  Interventions: Biological: AAV RPE65

INTERVENTIONS:
Biological: AAV RPE65 — Comparison of different dosages of AAV RPE65

SUMMARY:
A clinical trial of AAV2/5 vector for patients with Defects in RPE65

DETAILED DESCRIPTION:
A dose escalation and dose expansion (Phase I/II) trial of adults and children with retinal dystrophy associated with defects in RPE65. ATIMP will be administered to one eye only in a single sub-retinal procedure

ELIGIBILITY:
Key Inclusion Criteria:

* Aged 3 years or older
* Early-onset severe retinal dystrophy consistent with RPE65 deficiency

Key Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Have participated in another research study involving an investigational therapy for ocular disease within the last 6 months.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-04; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Kellogg Eye Centre, University of Michigan, Ann Arbor, Michigan, United States
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose AAV-RPE65: Unilateral sub-retinal injection of AAV2/5-OPTIRPE65 in a total volume of no more than 1mL at low dose (1 x 10^11 vg/mL)
- Intermediate Dose AAV-RPE65: Unilateral sub-retinal injection of AAV2/5-OPTIRPE65 in a total volume of no more than 1mL at intermediate dose (3 x 10^11 vg/mL)
- High Dose AAV-RPE65: Unilateral sub-retinal injection of AAV2/5-OPTIRPE65 in a total volume of no more than 1mL at high dose (1 x 10^12 vg/mL)
Period: Overall Study
Arm/Group | Low Dose AAV-RPE65 | Intermediate Dose AAV-RPE65 | High Dose AAV-RPE65
Started | 9 | 3 | 3
Completed | 9 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose AAV-RPE65 | Intermediate Dose AAV-RPE65 | High Dose AAV-RPE65 | Total
Number analyzed (Participants) | 9 | 3 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.8 (5.52) | 19.0 (2.65) | 21.0 (3.00) | 15.7 (5.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 0 | 9
  Male | 2 | 1 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 2 | 3 | 14
  Black or African American | 0 | 0 | 1 | 1
  Asian | 2 | 0 | 0 | 2
  White | 7 | 3 | 2 | 12
Region of Enrollment [Number; unit: participants]
  United States | 2 | 0 | 0 | 2
  United Kingdom | 7 | 3 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Overall Safety of Adeno-Associated Virus Vector (AAV-OPTIRPE65) - Number of Participants With a Safety Event
Description: Safety was defined as an advanced therapy investigational medicinal product (ATIMP) related:
  * Reduction in visual acuity by 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters or more.
  * Severe unresponsive inflammation.
  * Infective endophthalmitis.
  * Ocular malignancy.
  * Grade III or above non-ocular suspected unexpected serious adverse reaction (SUSAR).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose AAV-RPE65 | Intermediate Dose AAV-RPE65 | High Dose AAV-RPE65
Number analyzed (Participants) | 9 | 3 | 3
Participants
  Number of subjects with dose limiting events. | 0 | 0 | 1
  Reduction in visual acuity by 15 ETDRS | 0 | 0 | 1
  Severe unresponsive inflammation | 0 | 0 | 0
  Infective endophthalmitis | 0 | 0 | 0
  Ocular malignancy | 0 | 0 | 0
  Grade III or above non-ocular SUSAR | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Within 6 months of ATIMP administration.
Description: A serious adverse event that started on or after the start of the administration of ATIMP. Any serious adverse events that occurred after the last administration of ATIMP + 6 months were not considered treatment emergent.
Arm/Group | Low Dose AAV-RPE65 | Intermediate Dose AAV-RPE65 | High Dose AAV-RPE65
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/9 | 2/3 | 1/3
Other Adverse Events (participants affected / at risk) | 5/9 | 2/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose AAV-RPE65 (N=9) | Intermediate Dose AAV-RPE65 (N=3) | High Dose AAV-RPE65 (N=3)
Uveitis (Eye disorders) | 0 (0) | 2 (2) | 1 (1) — ATIMP Related
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — ATIMP Related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose AAV-RPE65 (N=9) | Intermediate Dose AAV-RPE65 (N=3) | High Dose AAV-RPE65 (N=3)
Uveitis (Eye disorders) | 3 (3) | 1 (1) | 1 (2) — ATIMP Related
Visual acuity reduced (Eye disorders) | 2 (2) | 0 (0) | 1 (1) — ATIMP Related
Anterior chamber inflammation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — ATIMP Related
Hypotony of eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — ATIMP Related
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — ATIMP Related
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) — ATIMP Related
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — ATIMP Related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT02781480/Prot_SAP_000.pdf